CLINICAL TRIAL: NCT01625429
Title: A Single-center, Prospective, Phase II Study of Albumin-bound Paclitaxel (Nab-paclitaxel) and Carboplatin With or Without Trastuzumab (Herceptin) as Neoadjuvant Therapy in Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Study of Nab-paclitaxel Plus Carboplatin in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX-1201
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neoadjuvant (Experimental)
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel 125mg/m2, day 1, 8, 15, q4w; carboplatin AUC 2, day 1, 8, 15, q4w; for HER-2 positive patients: trastuzumab loading dose 4mg/kg, then 2mg/kg, day 1, 8, 15, 22, q4w. All patients will receive up to four cycles except for unacceptable toxicity
  Other Names: Abraxane; Herceptin

SUMMARY:
This is a single-center, prospective, single arm phase II study to evaluate the efficacy and safety of nab-paclitaxel plus carboplatin (with trastuzumab for HER-2 positive patients) as neoadjuvant therapy in operable locally advanced breast cancer patients. The primary objective is pCR. The secondary objectives include ORR, 3-yr DFS, OS and safety. The sample size is 30.

ELIGIBILITY:
Inclusion Criteria:

* Female, between 18 and 70 years old
* Life expectancy is more than 12 months
* Breast MRI or ultrasound confirmd tumor over 3cm and biopsy comfirned invasive breast caner of stage II-III (inflammatory breast cancer excluded)
* Not accompanied with other malignancies（except for controlled carcinoma in situ of the cervix or skin basal-cell carcinoma）
* A normal bone marrow: absolute neutrophil count≥1.5*10E9/L, hemoglobin≥100g/L, PLT≥100*10E9/L
* Normal liver and renal functions: AST≤60U/L, total biliruin≤1.5*upper limit of normal, serum creatinine≤110umol/L, urea nitrogen≤7.1mmol/L
* Normal blood coagulation function
* ECOG performance status of 0-1
* Willing to coordinate with a punch biopsy before treatment and accept neoadjuvant therapy
* Women of child-producing potential must agree to use effective contraceptive methods during the study, and a negative serum or urine pregnancy test must be obtained within 7 days prior to administration of the drugs
* Written informed consent
* For HER-2 positive patients, the HER-2 status must be determined by ICH +++ or FISH/CISH. For patients treated with trastuzumb, LVEF≥55% by ultrasonic cardiogram or MUGA scan

Exclusion Criteria:

* Previous systematic or local therapy including chemotherapy for breast cancer
* Distant metastases of breast cancer are observed
* Concurrent uncontrolled lung disease, severe sepsis, active peptic ulcer requring treatment, blood coagulation disorders, serious uncontrolled diabetes, connective tissue disease or bone marrow depression, unable to tolerate neoadjuvant therapy and related treatment
* >Grade 1 peripheral neuropathy caused by any reason
* History of CHF, uncontrolled symptomatic angina, history of arrhythmias or myocardial infarction, poorly controlled hypertension (systolic pressure > 180mmHg or diastlic pressure > 100 mmHg)
* Lactational or gestational breast cancer
* Not willing to accept a punch biopsy before treatment and neoadjuvant therapy
* Psychopath or any other reasons that would preclude compliane with treatment
* Known serious allergy to any of the study drugs or excipients
* Participation in another study requiring administration of an in investigational drug or biological agent at present or recently (within the last 30 days prior to screening visit)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | Obtained within six months of the last patient's enrollment
  The percentage of patients with a pathological complete response after neoadjuvant therapy

SECONDARY OUTCOMES:
Overall response rate | Obtained within six months of the last patient's enrollment
  The percentage of patients with complete response or partial response after neoadjuvant therapy
Three-year disease free survival | Obtained within 42 months after last patient's enrollment
  The percentage of patients who survive without breast cancer recurrence or metastases three years after surgery
Overall survival | Obtained around 5 years after the last patient's erollment
  The overall survival time of all patients enrolled in the study presented by survival curve and median value
Safety | Obtained around six months after the last patient's enrollment
  List and frequencies of adverse events occured during and one-month after the investigational drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China